CLINICAL TRIAL: NCT03368144
Title: Belgian Prospective, Non-randomized Multi-center, Controlled Physician-initiated Trial: Evaluation of the Safety and Efficacy of the ClearLumen II Peripheral Thrombectomy System Recanalization of Acute and Subacute Thrombotic Femoropopliteal Occlusions
Brief Title: Belgian Trial Evaluating the ClearLumen II Peripheral Thrombectomy System Recanalization of (sub)acute Thrombotic Femoropopliteal Occlusions
Acronym: BELTHROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BELTHROM-20170628
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ClearLumen II Peripheral Thrombectomy System (Experimental): Patients treated with the ClearLumen II Peripheral Thrombectomy System
  Interventions: Device: ClearLumen II Peripheral Thrombectomy System

INTERVENTIONS:
Device: ClearLumen II Peripheral Thrombectomy System — Patients will be treated with the ClearLumen Peripheral Stent Graft System

SUMMARY:
The BELTHROM trial investigates the efficacy and safety of the ClearLumen II Peripheral Thrombectomy System recanalization of acute and subacute thrombotic femoropopliteal occlusions (Acute Limb Ischemia (ALI); Rutherford I, IIa, IIb and III). An expected total of 50 patients will be treated. The lesion is located within the femoropopliteal artery (native, in-stent or bypass graft). During the procedure, the device is introduced, activated and slowly advanced into the occlusion to clean out the wall-adherent thrombotic material. If residual underlying stenosis of >30% persists additional endovascular treatment can be performed according to the physician's discretion. Patients will be invited for a follow-up visit at 1 month post-procedure. The primary efficacy endpoint is the technical success of the ClearLumen II Peripheral Thrombectomy System, defined as removal of ≥90% acute clot as documented by angiography. The primary safety endpoint is defined as the absence of device-related complications, which is defined as embolization, perforation or dissection caused by the ClearLumen II Peripheral Thrombectomy System. Secondary endpoints include procedural success, percent clot removed by the ClearLumen II Peripheral Thrombectomy System, clinical success at 1 month follow-up visit, 30-day target lesion revascularization, 30-days serious adverse events and 30-days adverse events.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to evaluate, in a controlled setting, the safety and efficacy of the recanalization of acute and subacute thrombotic (up to 6 weeks) femoropopliteal occlusions with the ClearLumen II Peripheral Thrombectomy System.

Patients will be selected based on the investigator's assessment, evaluation of the underlying disease and the eligibility criteria. The patient's medical condition should be stable, with no underlying medical condition which would prevent them from performing the required testing or from completing the study. Patients should also be geographically stable, willing and able to cooperate in this clinical study and remain available for follow-up. A patient is considered enrolled in the study after obtaining the patients informed consent, if there is full compliance with the study eligibility criteria and after successful guidewire passage through the study target lesion.

Prior to the index procedure the following tests and clinical data will be collected: informed consent for data collection, demographics, medical history, medication record, physical examination, clinical category of acute limb ischemia (Rutherford category) and resting ankle-brachial index (ABI).

During the procedure, the occlusion needs first to be recanalized by conventional guidewire technique, since the ClearLumen II Peripheral Thrombectomy System is an over-the-wire system (0.035"). After assessment of the lesion by angiography via a common femoral artery approach (contralateral/ipsilateral) the occlusion is intraluminally crossed with the wire according to physician's discretion. Afterwards, the device is introduced and the catheter is activated. Then the catheter is slowly advances into the occlusion. Several passages of the occlusion may needed to clean out all wall-adherent thrombotic material. If residual underlying stenosis of >30% persists additional endovascular treatment can be performed according to the physician's discretion.

The regular follow-up is necessary to monitor the condition of the patient and the result of the procedure. Patients will be invited for a follow-up visit 1 month after the index procedure. The following data will be collected during this follow-up visit: medication record, physical examination, rutherford categorization, ABI and color flow doppler ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Presence of acute (less than 14 days) or subacute (2-6 weeks) limb ischemia or acute femoropopliteal thrombus during a revascularization procedure (native, in-stent or bypass graft) (acute limb ischemia (ALI) Rutherford I, IIa, IIb, III)
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient is candidate for thrombolytic, anticoagulation or antiplatelet therapy
* Target vessel diameter ≥ 3 mm

Exclusion Criteria:

* Chronic total occlusion of the target segment
* Absence of at least one continuous patent runoff vessel to the foot
* Inability to cross the lesion with a guidewire
* Known bacteremia at the time of intervention
* Untreated flow-limiting inflow lesions
* Aneurysm in the target vessel
* Visual stent deformations/fractures
* Severe medical comorbidities (untreated coronary artery disease/congestive heart failure, severe chronic obstructive pulmonary disease, metastatic malignancy, dementia, etc) limiting life expectancy to < 6 months or other medical condition that in the opinion of the investigator would prelude compliance with the study protocol
* Presence of gangrene or osteomyelitis
* Any previously known coagulation disorder, including hypercoagulability
* Contraindication to anticoagulation or antiplatelet therapy
* Patient with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Technical success | During index procedure
  Removal of ≥90% acute clot as documented by angiography
Primary safety endpoint | During index procedure
  Absence of device-related complications

SECONDARY OUTCOMES:
Procedural success | During index procedure
  Re-establishment of flow in the target segment with residual stenosis ≤30% using any adjunctive technique as deemed necessary by the investigator
Target Lesion Revascularization (TLR) | 30 days post-procedure
  Repeated intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge
Clinical success | 30 days post-procedure
  Improvement of Rutherford classification of one or more classes as compared to the pre-procedure Rutherford classification
Serious adverse events (SAEs) | 30 days post-procedure
  Death, stroke, myocard infarction, unplanned major amputation or any clinical life threatening event
Adverse events (AEs) | 30 days post-procedure
  Any clinical event requiring escalation of therapy or prolonging of the hospitalization as judged by the investigator
2nd efficacy endpoint | During index procedure
  Percent clot removed by the ClearLumen II Peripheral Thrombectomy System

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Study Director — ID3 Medical
Locations (3):
- Belgium (3):
  - O.L.V. Hospital, Aalst
  - A.Z. Sint-Blasius, Dendermonde
  - Z.O.L., Genk